CLINICAL TRIAL: NCT00531479
Title: A Prospective, Randomized Trial Comparing The Efficacy Of Anidulafungin And Voriconazole In Combination To That Of Voriconazole Alone When Used For Primary Therapy Of Proven Or Probable Invasive Aspergillosis
Brief Title: Anidulafungin Plus Voriconazole Versus Voriconazole For The Treatment Of Invasive Aspergillosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8851009
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole; Anidulafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voriconazole (Active Comparator): Voriconazole monotherapy
  Interventions: Drug: voriconazole
- Voriconazole and Anidulafungin (Experimental): Combination therapy with voriconazole and anidulafungin
  Interventions: Drug: anidulafungin; Drug: voriconazole

INTERVENTIONS:
Drug: voriconazole — First week: Voriconazole 6 mg/kg IV bid for the first 24 hours, followed by 4 mg/kg IV BID plus anidulafungin placebo IV qd.
  Second week: Voriconazole 4 mg/kg IV bid or 300 mg PO bid plus anidulafungin placebo IV qd.
  Third and fourth weeks: Voriconazole 4 mg/kg IV bid OR 300 mg PO bid plus anidulafungin placebo IV qd,
  OR
  Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Fifth and sixth weeks: Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Other Names: Vfend
  Arms: Voriconazole
Drug: anidulafungin — First week: Voriconazole 6 mg/kg IV bid for the first 24 hours, followed by 4 mg/kg IV bid plus anidulafungin 200 mg IV on day 1, followed by 100 mg IV qd thereafter.
  Second week: Voriconazole 4 mg/kg IV bid or 300 mg PO bid plus anidulafungin 100 mg IV qd.
  Third and fourth weeks: Voriconazole 4 mg/kg IV bid OR 300 mg PO bid plus anidulafungin 100 mg IV qd,
  OR
  Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Fifth and sixth weeks: Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Other Names: Eraxis
  Arms: Voriconazole and Anidulafungin
Drug: voriconazole — First week: Voriconazole 6 mg/kg IV bid for the first 24 hours, followed by 4 mg/kg IV bid plus anidulafungin 200 mg IV on day 1, followed by 100 mg IV qd thereafter.
  Second week: Voriconazole 4 mg/kg IV bid or 300 mg PO bid plus anidulafungin 100 mg IV qd.
  Third and fourth weeks: Voriconazole 4 mg/kg IV bid OR 300 mg PO bid plus anidulafungin 100 mg IV qd,
  OR
  Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Fifth and sixth weeks: Voriconazole 4 mg/kg IV bid or 300 mg PO bid monotherapy.
  Other Names: Vfend
  Arms: Voriconazole and Anidulafungin

SUMMARY:
This study compares the effectiveness and safety of the combination of anidulafungin and voriconazole compared to that of voriconazole alone (which is generally considered the standard of care) for the treatment of Invasive Aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised state due to either 1. receipt of hematopoeitic stem cell transplantation or 2. hematologic malignancy;
* Diagnosis of possible, probable, or proven invasive aspergillosis.

Exclusion Criteria:

* Patients with aspergilloma or chronic aspergillosis
* Receipt of 4 or more days of systemic antifungal treatment for the current episode of invasive aspergillosis
* Anticipated survival of less than 5 days or Karnofsky score <=20

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (18):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Seattle, Washington
- Australia (3):
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
- Belgium (4):
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Yvoir
- Brazil (3):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Rio de Janeiro, Rio de Janeiro
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
- Canada (4):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Hamilton, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, Prague, Czechia
- France (8):
  - Pfizer Investigational Site, Nantes, Cedex 01
  - Pfizer Investigational Site, Marseille, Cedex 09
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Créteil
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Strasbourg
- Germany (11):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Cologne
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Frankfurt (Oder)
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg/Saar
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Würzburg
- Pfizer Investigational Site, Thessaloniki, Greece
- Pfizer Investigational Site, Pune, Maharashtra, India
- Italy (6):
  - Pfizer Investigational Site, Cuneo
  - Pfizer Investigational Site, Genova
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Pescara
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, RC Leiden, Netherlands
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Poland (2):
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Warsaw
- Pfizer Investigational Site, Lisbon, Portugal
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Saint Petersburg
- Pfizer Investigational Site, Singapore, Singapore, Singapore
- Pfizer Investigational Site, Seoul, South Korea
- Spain (4):
  - Pfizer Investigational Site, Badalona, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Salamanca, Salamanca
  - Pfizer Investigational Site, Valencia, Valencia
- Switzerland (2):
  - Pfizer Investigational Site, Geneva
  - Pfizer Investigational Site, Lausanne
- Taiwan (3):
  - Pfizer Investigational Site, Kuei-Shan Hsiang, Taoyuan County
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei
- Thailand (2):
  - Pfizer Investigational Site, Bangkok, Thailand
  - Pfizer Investigational Site, Bangkok
- Turkey (Türkiye) (2):
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Ankara
- United Kingdom (2):
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- [Derived] Marr KA, Schlamm HT, Herbrecht R, Rottinghaus ST, Bow EJ, Cornely OA, Heinz WJ, Jagannatha S, Koh LP, Kontoyiannis DP, Lee DG, Nucci M, Pappas PG, Slavin MA, Queiroz-Telles F, Selleslag D, Walsh TJ, Wingard JR, Maertens JA. Combination antifungal therapy for invasive aspergillosis: a randomized trial. Ann Intern Med. 2015 Jan 20;162(2):81-9. doi: 10.7326/M13-2508. PMID 25599346
- [Derived] Liu P, Mould DR. Population pharmacokinetic-pharmacodynamic analysis of voriconazole and anidulafungin in adult patients with invasive aspergillosis. Antimicrob Agents Chemother. 2014 Aug;58(8):4727-36. doi: 10.1128/AAC.02809-13. Epub 2014 Jun 9. PMID 24914120
- [Derived] Liu P, Mould DR. Population pharmacokinetic analysis of voriconazole and anidulafungin in adult patients with invasive aspergillosis. Antimicrob Agents Chemother. 2014 Aug;58(8):4718-26. doi: 10.1128/AAC.02808-13. Epub 2014 Jun 9. PMID 24913161
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851009&StudyName=Anidulafungin%20Plus%20Voriconazole%20versus%20Voriconazole%20For%20The%20Treatment%20Of%20Invasive%20Aspergillosis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified at study entry for host and transplant variables known to have an independent impact on the probablity of death due to invasive aspergillosis (IA) (allogenic hematopoietic stem cell transplant versus other, and pulmonary IA).
Groups:
- Voriconazole/Anidulafungin: Week 1: Voriconazole 6 mg/kg intravenously (IV) twice a day (bid) for 24 hours, followed by voriconazole 4 milligrams per kilogram (mg/kg) IV BID plus anidulafungin 200 mg IV on day 1, followed by 100 mg IV once a day (QD); Week 2: Voriconazole 4 mg/kg IV BID or 300 mg orally (PO) BID plus anidulafungin 100 mg IV QD; Weeks 3 and 4: voriconazole 4 mg/kg IV BID or 300 mg PO BID plus anidulafungin 100 mg IV QD or voriconazole 4 mg/kg IV BID or 300 mg PO BID monotherapy; Weeks 5 and 6: voriconazole 4 mg/kg IV BID or 300 mg PO BID monotherapy.
- Voriconazole / Placebo: Week 1: Voriconazole 6 mg/kg IV BID for 24 hours, followed by voriconazole 4 mg/kg IV BID plus anidulafungin placebo IV QD; Week 2: voriconazole 4 mg/kg IV BID or voriconazole 300 mg PO BID plus anidulafungin placebo IV QD through Day 14; Weeks 3 and 4: voriconazole 4 mg/kg IV BID or 300 mg PO BID plus anidulafungin placebo; Weeks 5 and 6: voriconazole 4 mg/kg IV BID or 300 mg PO BID monotherapy.
Period: Overall Study
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Started | 230 | 229
Treated | 228 | 226
Completed | 154 | 146
Not Completed | 76 | 83
Not completed — Death | 68 | 71
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Did not receive treatment | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo | Total
Number analyzed (Participants) | 228 | 226 | 454
Age Continuous [Mean (Standard Deviation); unit: years] | 52.0 (15.4) | 51.0 (15.9) | 51.5 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 95 | 189
  Male | 134 | 131 | 265

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality at Week 6 in Participants With Proven or Probable Invasive Aspergillosis
Description: Number of deaths measured 6 weeks after start of treatment. Time to death defined as date of death minus first treatment date + 1.
Time Frame: Day 1 to Day 42 (Week 6)
Population: Modified intent-to-treat (MITT) population: all randomized participants with proven or probable IA confirmed by Day 7 following enrollment who received at least 1 dose of study medication. N=number of participants in MITT population at Week 6. Participants not known to have died were censored at last study visit (Day 84).
Measure: Number; unit: participants
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
participants | 26 | 39
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; All-cause mortality calculated using the Kaplan-Meier (KM) product limit estimator on Day 42 (Week 6) within each stratum and weighted by the harmonic mean of the sample sizes in the strata. Treatment difference (stratified) based on a weighted difference in proportions. Stratification variables were site of infection and host factors; Test type: Superiority or Other; p = 0.0434, Z test for difference in proportions — P-value based on a 1-sided test and tested against a 1-sided alpha of 0.025 to determine statistical significance; Mean Difference (Final Values) = -8.74, 95% CI 2-sided [-18.99 to 1.51] — The 95% CI was based on using Greenwood's formula for the variance of the KM estimator

2. Secondary Outcome: Global Response at Week 6
Description: Number of participants with a successful response (complete or partial global response). Complete response = resolution of all clinical signs and symptoms and >90% of lesions due to IA that were visible on radiologic studies at baseline (BL); partial response = clinical improvement and >50% improvement in radiological findings present at BL.
Time Frame: Baseline, Day 42 (Week 6)
Population: MITT; N = number of participants in MITT population at Week 6. Missing data and participants who died at Week 6 were treated as failure.
Measure: Number; unit: participants
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
participants | 44 | 61
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; Treatment difference (stratified) based on a weighted difference in proportions. Stratification variables: site of infection and host factors; Test type: Superiority or Other; P-value for global response was to be reported only if Week 6 mortality was significant; Mean Difference (Final Values) = -10.23, 95% CI 2-sided [-21.6 to 1.15] — 95% confidence interval based on the difference in success rates using the normal approximation to the binoial distribution

3. Secondary Outcome: All-cause Mortality at Week 6 in Participants With Possible, Probable, or Proven Invasive Aspergillosis (IA)
Description: Number of deaths due to any cause measured 6 weeks after start of treatment. Time to death defined as date of death minus first treatment date + 1.
Time Frame: Day 1 to Day 42 (Week 6)
Population: Intent-to-treat (ITT) population: participants in MITT analysis set plus participants with possible IA who could not be upgraded to probable or proven IA within 7 days and had received at least 1 dose of study medication. N=number of participants in ITT population at Week 6.
Measure: Number; unit: participants
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 215 | 207
participants | 44 | 47
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2611, Z test for difference in proportions — P-Value based on a 1-sided test and tested against a 1-sided alpha of 0.025 to determine statistical significance; Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-10.77 to 5.56] — 95% confidence interval based on using Greenwood's formula for the variance of the Kaplan Meier estimator

4. Secondary Outcome: All-cause Mortality at Week 12 in Participants With Probable or Proven Invasive Aspergillosis (IA)
Description: Number of deaths due to any cause measured 12 weeks after start of treatment. Time to death defined as date of death minus first treatment date + 1.
Time Frame: Day 1 to Day 84 (Week 12)
Population: MITT; N=number of participants in MITT population at Week 12.
Measure: Number; unit: participants
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
participants | 39 | 55
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0383, Z test for difference in proportions — P-Value based on a 1-sided test and tested against a 1-sided alpha of 0.025 to determine statistical significance; Mean Difference (Final Values) = -10.18, 95% CI 2-sided [-21.44 to 1.09] — 95% confidence intervalbased on using Greenwood's formula for the variance of the Kaplan Meier estimator

5. Secondary Outcome: Mortality Due to Invasive Aspergillosis (IA) at Week 6 in Participants With Probable or Proven IA
Description: Number of deaths due to Invasive Aspergillosis measured 6 weeks after start of treatment. Time to death defined as date of death minus first treatment date + 1.
Time Frame: Day 1 to Day 42 (Week 6)
Population: MITT; N = number of participants in MITT population at Week 6. Participants who died due to causes other than IA before Week 6 were censored at their time of death in this analysis.
Measure: Number; unit: participants
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
participants | 23 | 33
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1029, Z test for difference in proportions — P-Value based on a one-sided test and tested against a 1-sided alpha of 0.025 to determine statistical significance; Mean Difference (Final Values) = -6.24, 95% CI 2-sided [-15.9 to 3.42] — 95% confidence interval based on Greenwood's formula for the variance of the Kaplan Meier estimator

6. Secondary Outcome: Time to Death: All-Cause Mortality
Description: Survival time from start of treatment. Time to death defined as date of death due to any cause minus first treatment date + 1.
Time Frame: Day 1 to Day 84 (Week 12)
Population: MITT; N = number of participants in MITT population at time of assessment.
Measure: Median (Full Range); unit: days
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
days | 30.0 [2 to 84] | 30.0 [3 to 79]
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; Hazard Ratio: hazard of death in the Voriconazole/Anidulafungin arm relative to the Voriconazole/Placebo arm, adjusted for host factor status and site of infection. Participants who died beyond Day 84 were censored; Test type: Superiority or Other; p = 0.083, Cox proportional hazards model; Hazard Ratio (HR) = 0.696, 95% CI 2-sided [0.46 to 1.04]

7. Secondary Outcome: Time to Death Due to Invasive Aspergillosis (IA)
Description: Survival time from start of treatment. Time to death defined as date of death due to IA minus first treatment date + 1.
Time Frame: Day 1 to Day 84 (Week 12)
Population: MITT; N = number of participants in MITT population at time of assessment. Participants who died due to causes other than IA were defined as censored at time of death.
Measure: Median (Full Range); unit: days
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Number analyzed (Participants) | 135 | 142
days | 14.0 [2 to 40] | 18.5 [4 to 45]
Statistical Analysis 1: Comparison: Voriconazole/Anidulafungin vs Voriconazole / Placebo; Analysis based on Cox proportional hazards model. Participants who died beyond day 84 were censored; Test type: Superiority or Other; p = 0.164, Cox proportional hazards model; Hazard Ratio (HR) = 0.687, 95% CI 2-sided [0.40 to 1.16] — 95% confidence interval based on Greenwood's formula

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Voriconazole/Anidulafungin | Voriconazole / Placebo
Serious Adverse Events (participants affected / at risk) | 115/228 | 104/226
Other Adverse Events (participants affected / at risk) | 194/228 | 192/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole/Anidulafungin (N=228) | Voriconazole / Placebo (N=226)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Blood disorder (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileitis (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Disease progression (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 2
Multi-organ failure (General disorders) | 5 | 4
Pyrexia (General disorders) | 3 | 4
Sudden cardiac death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 2
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatic vein occlusion (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 1
Aspergillosis (Infections and infestations) | 6 | 5
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Hepatic infection fungal (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Meningitis fungal (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 5
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 9 | 7
Septic shock (Infections and infestations) | 10 | 14
Sinusitis (Infections and infestations) | 0 | 1
Sinusitis aspergillus (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Streptococcal sepsis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Zygomycosis (Infections and infestations) | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1
Cytomegalovirus test positive (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Procalcitonin increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia plasmacytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 2
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 2
Epilepsy (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Toxic neuropathy (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephritic syndrome (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 5 | 0
Renal impairment (Renal and urinary disorders) | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Iliac artery thrombosis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole/Anidulafungin (N=228) | Voriconazole / Placebo (N=226)
Anaemia (Blood and lymphatic system disorders) | 7 | 13
Tachycardia (Cardiac disorders) | 12 | 19
Vision blurred (Eye disorders) | 14 | 11
Abdominal pain (Gastrointestinal disorders) | 14 | 12
Abdominal pain upper (Gastrointestinal disorders) | 9 | 15
Constipation (Gastrointestinal disorders) | 35 | 30
Diarrhoea (Gastrointestinal disorders) | 39 | 37
Dyspepsia (Gastrointestinal disorders) | 6 | 12
Nausea (Gastrointestinal disorders) | 38 | 42
Vomiting (Gastrointestinal disorders) | 32 | 23
Chest pain (General disorders) | 16 | 9
Chills (General disorders) | 13 | 10
Fatigue (General disorders) | 5 | 14
Mucosal inflammation (General disorders) | 10 | 15
Oedema (General disorders) | 12 | 14
Oedema peripheral (General disorders) | 34 | 34
Pain (General disorders) | 10 | 13
Pyrexia (General disorders) | 28 | 42
Fall (Injury, poisoning and procedural complications) | 12 | 4
Aspartate aminotransferase increased (Investigations) | 12 | 13
Blood alkaline phosphatase increased (Investigations) | 20 | 6
Decreased appetite (Metabolism and nutrition disorders) | 15 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 30
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 11
Headache (Nervous system disorders) | 16 | 26
Agitation (Psychiatric disorders) | 13 | 7
Anxiety (Psychiatric disorders) | 12 | 15
Confusional state (Psychiatric disorders) | 10 | 15
Hallucination, visual (Psychiatric disorders) | 7 | 12
Insomnia (Psychiatric disorders) | 29 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 20
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 12
Rash (Skin and subcutaneous tissue disorders) | 30 | 31
Hypertension (Vascular disorders) | 32 | 21
Hypotension (Vascular disorders) | 30 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.